CLINICAL TRIAL: NCT04822142
Title: Congenital Cytomegalovirus Infection in Vietnam: Prevalence, Morbidity and Risk Factors
Brief Title: Congenital CYtoMEgalovirus Infection in VIEtnam (CYMEVIE)
Acronym: CYMEVIE
Status: Recruiting | Type: Observational
Sponsor: Hanoi Obstetrics and Gynecology Hospital (Other)
Collaborators: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Sponsor
Other Study IDs: PSHN.0003.2021
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Prenatal Infection; Congenital Infection; Neonatal Disease
Keywords: CYMEVIE; Cytomegalovirus; Congenital Cytomegalovirus infection; CMV PCR; CMV; cCMV
MeSH Terms: conditions — Infant, Newborn, Diseases; Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Maternal whole blood, saliva and urine collected in the first trimester of pregnancy. Maternal whole blood and urine collected at time of delivery. Neonatal saliva sample collected within 72 hours after birth. Heel-prick blood sample on paper within 72 hours after birth. For neonates with positive CMV PCR on saliva sample, neonatal urine during first month will be collected, whole blood at moment of 1st month follow-up will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To estimate the prevalence of congenital CMV infection in Vietnamese neonates and relating morbidity within 2-year follow-up. Along with evaluating the predictive value of the presence and the level of CMV replication in the first trimester in a highly seropositive population

DETAILED DESCRIPTION:
Congenital cytomegalovirus infection (cCMV) is the main non-genetic cause of sensorineural hearing loss (SNHL), and a major cause of neuro-disability. High maternal CMV prevalence seems to be consistently associated with high prevalence of cCMV infection but the associated morbidity might be different from one population to another.

There exists no serologic marker useful to differentiate non-primary infection from primary infection. Since the morbidity of cCMV is similar between both primary and non-primary maternal infection, and to be infected in the first trimester is the major risk factor for long-term sequelae in neonates. Hence, it is needed to focus on finding markers that predict cCMV after maternal infection in the first trimester of pregnancy.

To date, the epidemiology of cCMV, the morbidity related to cCMV in Vietnamese population and the predictive value of Cytomegalovirus Polymerase Chain Reaction (CMV PCR) in maternal blood and urine in the first trimester remain unknown. Therefore, it is necessary to conduct this study.

ELIGIBILITY:
Inclusion Criteria:

* Vietnamese pregnant women in the first trimester of pregnancy and at delivery and subsequent live neonates at birth.
* Informed consent

Exclusion Criteria:

* Women under 18 years old.
* Miscarriages
* Stillbirths
* Premature delivery before 34th gestational week
* Loss to follow-up maternal monitoring.
* Participation in another interventional study that influences management of labour at delivery or perinatal morbidity or mortality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 5,000 mother/neonate pairs
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of congenital CMV infection in Vietnamese neonates | Within 7 days from birth
  Number of CMV positive neonates among all tested neonates

SECONDARY OUTCOMES:
To estimate the prevalence of symptomatic cCMV in neonates | Up to 25 months from recruitment
  Proportion of neonates presenting with at least one symptom related to cCMV in all cCMV neonates
To estimate the prevalence of cCMV related hearing loss in neonates | Up to 25 months from recruitment
  Proportion of cCMV related hearing loss in neonates in all cCMV neonates
To estimate the prevalence of cCMV related neurological sequelae in neonates | Up to 25 months from recruitment
  Proportion of cCMV related neurological sequelae in neonates in all cCMV neonates
To estimate CMV seroprevalence in pregnant Vietnamese women | Up to 25 months from recruitment
  Proportion of seropositive women in all tested pregnant women, including mother of CMV positive neonates and control group
To evaluate the value of a positive CMV PCR in maternal whole blood in the first trimester to predict infection in the neonates | Up to 25 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal whole blood in the first trimester between women who gave birth to an infected neonate and women gave birth to an uninfected neonate from control group
To evaluate the value of a positive CMV PCR in maternal urine in the first trimester to predict infection in the neonates | Up to 25 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal urine in the first trimester between women who gave birth to an infected neonate and women gave birth to an uninfected neonate from control group
To evaluate the value of a positive CMV PCR in maternal saliva in the first trimester to predict cCMV infection in the neonates | Up to 25 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal saliva in the first trimester between women who gave birth to an infected neonate and women gave birth to an uninfected neonate from control group
To evaluate the value of a positive CMV PCR in maternal whole blood at delivery to predict infection in the neonates | Up to 25 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal whole blood at delivery between women who gave birth to an infected neonate and women gave birth to an uninfected neonate from control group
To evaluate the value of a positive CMV PCR in maternal urine at delivery to predict infection in the neonates | Up to 25 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal urine at delivery between women who gave birth to an infected neonate and women gave birth to an uninfected neonate from control group
To evaluate the value of a positive CMV PCR in whole blood in the first trimester to predict the presence of symptomatic cCMV infection in neonates | Up to 25 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal whole blood in the first trimester between symptomatic infected neonates and asymptomatic infected neonates
To evaluate the value of a positive CMV PCR in maternal urine in the first trimester to predict a cCMV symptomatic infection in neonates | Up to 25 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal urine in the first trimester between symptomatic infected neonates and asymptomatic infected neonates
To evaluate the value of a positive CMV PCR in maternal saliva in the first trimester to predict the presence of symptomatic cCMV infection in neonates | Up to 25 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal saliva in the first trimester between symptomatic infected neonates and asymptomatic infected neonates
To evaluate the value of a positive CMV PCR in maternal whole blood at delivery to predict the presence of symptomatic cCMV infection in neonates | Up to 25 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal whole blood at delivery between symptomatic infected neonates and asymptomatic infected neonates
To evaluate the value of a positive CMV PCR in maternal urine at delivery to predict a cCMV symptomatic infection in neonates | Up to 25 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal urine at delivery between symptomatic infected neonates and asymptomatic infected neonates
To evaluate the association between CMV PCR viral load in maternal whole blood at first trimester and at delivery in mothers with infected neonates | Up to 25 months from recruitment
  Evaluation the change of CMV PCR viral load in maternal whole blood at first trimester and at delivery in mothers with infected neonates
To evaluate the association between CMV PCR viral load in maternal urine at first trimester and at delivery in mothers with infected neonates | Up to 25 months from recruitment
  Evaluation the change of CMV PCR viral load in maternal urine at first trimester and at delivery in mothers with infected neonates
To evaluate the association between CMV PCR viral load in maternal whole blood at first trimester and at delivery in mothers with uninfected neonates in control group | Up to 25 months from recruitment
  Evaluation the change of CMV PCR viral load in maternal whole blood at first trimester and at delivery in mothers with uninfected neonates in control group
To evaluate the association between CMV PCR viral load in maternal urine at first trimester and at delivery in mothers with uninfected neonates in control group | Up to 25 months from recruitment
  Evaluation the change of CMV PCR viral load in maternal urine at first trimester and at delivery in mothers with uninfected neonates in control group
To calculate the false positive rate of CMV PCR on neonatal saliva versus on dry blood spot in screening congenital CMV infection | Up to 25 months from recruitment
  Calculation of the rate of positive CMV PCR on neonatal saliva with a negative result on CMV PCR on neonatal dry blood spot in all CMV positive on neonatal saliva
To calculate the false positive rate of CMV PCR on neonatal saliva versus on urine in screening congenital CMV infection | Up to 25 months from recruitment
  Calculation of the rate of positive CMV PCR on neonatal saliva with a negative result on CMV PCR on neonatal urine in all CMV positive on neonatal saliva
To evaluate risks factors for cCMV in Vietnamese women | Up to 25 months from recruitment
  Factors that may differ between mothers of uninfected neonates and mothers of infected ones regarding maternal age, parity, gestity, twin pregnancy, known health conditions including hypertension, diabetes, HIV, auto immune diseases and living conditions will be analyzed
To estimate the prevalence of symptomatic cCMV at 2 years of age | Up to 48 months from recruitment
  Proportion of infants presenting with at least one symptom related to cCMV at 2 years of age in all cCMV infants
To estimate the prevalence of cCMV related hearing loss at 2 years of age | Up to 48 months from recruitment
  Proportion of infants with cCMV related hearing loss at 2 years of age in all cCMV infants
To estimate the prevalence of cCMV related neurological sequelae at 2 years of age | Up to 48 months from recruitment
  Proportion of infants with cCMV related neurological sequelae at 2 years of age in all cCMV infants
To evaluate the value of a positive CMV PCR in maternal whole blood in the first trimester to predict the cCMV long-term sequelae at the age of 2 years | Up to 48 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal whole blood in the first trimester between infected infants with long-term sequelae at 2 years of age and infected infants without long-term sequelae at 2 years of age
To evaluate the value of a positive CMV PCR in maternal urine in the first trimester to predict the cCMV long-term sequelae at the age of 2 years | Up to 48 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal urine in the first trimester between between infected infants with long-term sequelae at 2 years of age and infected infants without long-term sequelae at 2 years of age
To evaluate the value of a positive CMV PCR in maternal saliva in the first trimester to predict the cCMV long-term sequelae at the age of 2 years | Up to 48 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal saliva in the first trimester between between infected infants with long-term sequelae at 2 years of age and infected infants without long-term sequelae at 2 years of age
To evaluate the value of a positive CMV PCR in maternal whole blood at delivery to predict the cCMV long-term sequelae at the age of 2 years | Up to 48 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal whole blood at delivery between between infected infants with long-term sequelae at 2 years of age and infected infants without long-term sequelae at 2 years of age
To evaluate the value of a positive CMV PCR in maternal urine at delivery to predict the cCMV long-term sequelae at the age of 2 years | Up to 48 months from recruitment
  Comparison of the proportion of a positive CMV PCR in maternal urine at delivery between between infected infants with long-term sequelae at 2 years of age and infected infants without long-term sequelae at 2 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Yves Ville, MD.PhD, Study Chair — Hôpital Necker-Enfants Malades; Marianne Leruez-Ville, MD.PhD, Study Director — Hôpital Necker-Enfants Malades; Anh Nguyen Duy, MD.PhD, Study Director — Hanoi Obstetrics and Gynecology Hospital; Ha Nguyen Thi Thu, MD.PhD, Principal Investigator — Hanoi Obstetrics and Gynecology Hospital; Linh Dinh Thuy, MD.PhD, Principal Investigator — Hanoi Obstetrics and Gynecology Hospital
Locations (1):
- Hanoi Obstetrics and Gynecology Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No
To be determined

REFERENCES:
- [Background] Kenneson A, Cannon MJ. Review and meta-analysis of the epidemiology of congenital cytomegalovirus (CMV) infection. Rev Med Virol. 2007 Jul-Aug;17(4):253-76. doi: 10.1002/rmv.535. PMID 17579921
- [Background] Leruez-Ville M, Magny JF, Couderc S, Pichon C, Parodi M, Bussieres L, Guilleminot T, Ghout I, Ville Y. Risk Factors for Congenital Cytomegalovirus Infection Following Primary and Nonprimary Maternal Infection: A Prospective Neonatal Screening Study Using Polymerase Chain Reaction in Saliva. Clin Infect Dis. 2017 Aug 1;65(3):398-404. doi: 10.1093/cid/cix337. PMID 28419213
- [Background] Puhakka L, Renko M, Helminen M, Peltola V, Heiskanen-Kosma T, Lappalainen M, Surcel HM, Lonnqvist T, Saxen H. Primary versus non-primary maternal cytomegalovirus infection as a cause of symptomatic congenital infection - register-based study from Finland. Infect Dis (Lond). 2017 Jun;49(6):445-453. doi: 10.1080/23744235.2017.1279344. Epub 2017 Jan 24. PMID 28116961
- [Background] Mussi-Pinhata MM, Yamamoto AY, Aragon DC, Duarte G, Fowler KB, Boppana S, Britt WJ. Seroconversion for Cytomegalovirus Infection During Pregnancy and Fetal Infection in a Highly Seropositive Population: "The BraCHS Study". J Infect Dis. 2018 Sep 8;218(8):1200-1204. doi: 10.1093/infdis/jiy321. PMID 29868783
- [Background] Ross SA, Fowler KB, Ashrith G, Stagno S, Britt WJ, Pass RF, Boppana SB. Hearing loss in children with congenital cytomegalovirus infection born to mothers with preexisting immunity. J Pediatr. 2006 Mar;148(3):332-6. doi: 10.1016/j.jpeds.2005.09.003. PMID 16615962
- [Background] Yamamoto AY, Anastasio ART, Massuda ET, Isaac ML, Manfredi AKS, Cavalcante JMS, Carnevale-Silva A, Fowler KB, Boppana SB, Britt WJ, Mussi-Pinhata MM. Contribution of Congenital Cytomegalovirus Infection to Permanent Hearing Loss in a Highly Seropositive Population: The Brazilian Cytomegalovirus Hearing and Maternal Secondary Infection Study. Clin Infect Dis. 2020 Mar 17;70(7):1379-1384. doi: 10.1093/cid/ciz413. PMID 31102409
- [Background] Wang S, Wang T, Zhang W, Liu X, Wang X, Wang H, He X, Zhang S, Xu S, Yu Y, Jia X, Wang M, Xu A, Ma W, Amin MM, Bialek SR, Dollard SC, Wang C. Cohort study on maternal cytomegalovirus seroprevalence and prevalence and clinical manifestations of congenital infection in China. Medicine (Baltimore). 2017 Feb;96(5):e6007. doi: 10.1097/MD.0000000000006007. PMID 28151899
- [Background] Faure-Bardon V, Magny JF, Parodi M, Couderc S, Garcia P, Maillotte AM, Benard M, Pinquier D, Astruc D, Patural H, Pladys P, Parat S, Guillois B, Garenne A, Bussieres L, Guilleminot T, Stirnemann J, Ghout I, Ville Y, Leruez-Ville M. Sequelae of Congenital Cytomegalovirus Following Maternal Primary Infections Are Limited to Those Acquired in the First Trimester of Pregnancy. Clin Infect Dis. 2019 Oct 15;69(9):1526-1532. doi: 10.1093/cid/ciy1128. PMID 30596974